CLINICAL TRIAL: NCT02273297
Title: Exploring the Fuel-mediated Programming of Neonatal Growth
Brief Title: Healthy Start: Exploring the Fuel-mediated Programming of Neonatal Growth
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 09-0563; R01DK076648 (NIH); UL1TR001082 (NIH)
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy; Obesity
Keywords: Body composition; Body size
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women and their offspring: Ethnically diverse pregnant women and their offspring
  Interventions: Other: Maternal factors

INTERVENTIONS:
Other: Maternal factors

SUMMARY:
The purpose of this study is to establish and follow longitudinally a cohort of ethnically diverse pregnant women and their offspring, in order to explore the hypothesis that fetal over-nutrition is associated with obesity, metabolic, and cardiovascular abnormalities in the offspring.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women and infants
* Prior to 23 completed weeks of gestation
* Live in Colorado

Exclusion Criteria:

* Multiple gestation
* Preexisting

  * cancer
  * psychiatric disease
  * steroid-dependent asthma, or
  * diabetes
* Previous premature delivery prior to 25 weeks gestation or fetal demise

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants were recruited from prenatal obstetrics clinics at the University of Colorado Hospital outpatient pavilion.
Sampling Method: Non-Probability Sample
Enrollment: 2821 (Estimated)
Dates: Start 2009-07; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Fat mass | Birth
  Body composition assessed via air displacement plethysmography to calculate fat mass and fat-free mass.
Fat mass | 5 years
  Body composition assessed via air displacement plethysmography to calculate fat mass and fat-free mass.

SECONDARY OUTCOMES:
Fat mass | 5 months
  Body composition assessed via air displacement plethysmography to calculate fat mass and fat-free mass.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Dabelea, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Buck KE, Dhaliwal SK, Dabelea D, Perng W. Association of maternal psychosocial stress with newborn body composition in the Healthy Start study. J Dev Orig Health Dis. 2023 Oct;14(5):576-583. doi: 10.1017/S2040174423000223. Epub 2023 Sep 11. PMID 37694587
- [Derived] Dhaliwal SK, Dabelea D, Lee-Winn AE, Crume T, Wilkening G, Perng W. Maternal psychosocial stress during pregnancy and offspring neurobehavioral outcomes during early childhood in the Healthy Start Study. Ann Epidemiol. 2023 Oct;86:16-24.e3. doi: 10.1016/j.annepidem.2023.06.001. Epub 2023 Jun 14. PMID 37321280
- [Derived] Cohen CC, Harrall KK, Gilley SP, Perng W, Sauder KA, Scherzinger A, Shankar K, Sundaram SS, Glueck DH, Dabelea D. Body composition trajectories from birth to 5 years and hepatic fat in early childhood. Am J Clin Nutr. 2022 Oct 6;116(4):1010-1018. doi: 10.1093/ajcn/nqac168. PMID 36055960
- [Derived] Francis EC, Dabelea D, Boyle KE, Jansson T, Perng W. Maternal Diet Quality Is Associated with Placental Proteins in the Placental Insulin/Growth Factor, Environmental Stress, Inflammation, and mTOR Signaling Pathways: The Healthy Start ECHO Cohort. J Nutr. 2022 Mar 3;152(3):816-825. doi: 10.1093/jn/nxab403. PMID 34850052
- [Derived] Moore BF, Sauder KA, Starling AP, Hebert JR, Shivappa N, Ringham BM, Glueck DH, Dabelea D. Proinflammatory Diets during Pregnancy and Neonatal Adiposity in the Healthy Start Study. J Pediatr. 2018 Apr;195:121-127.e2. doi: 10.1016/j.jpeds.2017.10.030. Epub 2017 Dec 6. PMID 29217099
- [Derived] Perng W, Ringham BM, Glueck DH, Sauder KA, Starling AP, Belfort MB, Dabelea D. An observational cohort study of weight- and length-derived anthropometric indicators with body composition at birth and 5 mo: the Healthy Start study. Am J Clin Nutr. 2017 Aug;106(2):559-567. doi: 10.3945/ajcn.116.149617. Epub 2017 Jun 28. PMID 28659296
- [Derived] Boyle KE, Patinkin ZW, Shapiro AL, Baker PR 2nd, Dabelea D, Friedman JE. Mesenchymal Stem Cells From Infants Born to Obese Mothers Exhibit Greater Potential for Adipogenesis: The Healthy Start BabyBUMP Project. Diabetes. 2016 Mar;65(3):647-59. doi: 10.2337/db15-0849. Epub 2015 Dec 2. PMID 26631736
- [Derived] Starling AP, Brinton JT, Glueck DH, Shapiro AL, Harrod CS, Lynch AM, Siega-Riz AM, Dabelea D. Associations of maternal BMI and gestational weight gain with neonatal adiposity in the Healthy Start study. Am J Clin Nutr. 2015 Feb;101(2):302-9. doi: 10.3945/ajcn.114.094946. Epub 2014 Dec 3. PMID 25646327
- [Derived] Crume TL, Shapiro AL, Brinton JT, Glueck DH, Martinez M, Kohn M, Harrod C, Friedman JE, Dabelea D. Maternal fuels and metabolic measures during pregnancy and neonatal body composition: the healthy start study. J Clin Endocrinol Metab. 2015 Apr;100(4):1672-80. doi: 10.1210/jc.2014-2949. Epub 2015 Jan 9. PMID 25574704